CLINICAL TRIAL: NCT07014930
Title: Endobiotics for Phenotyping Cytochrome P450 Enzymes: Using Metabolomics to Identify Novel Endogenous CYP2C19 Activity Biomarkers in Healthy Volunteers
Brief Title: Identification of New Tools for Predicting Natural Metabolic Performance of the Liver
Acronym: Endo2C19
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Caroline Samer (Other)
Collaborators: Fonds national Suisse (Unknown)
Responsible Party: Sponsor-Investigator, Caroline Samer, Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-01956
Record Dates: First submitted 2025-05-19; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CYP2C19 Poor Metabolizers (PMs) (Experimental): Carriers of two non-functional alleles of CYP2C19
  Interventions: Drug: Control session; Drug: Inhibition session; Drug: Induction session
- CYP2C19 Normal, Rapid or Ultrarapid Metabolizers (NMs-RMs-UMs) (Experimental): Carriers of two normally functional alleles (NMs), one normally functional allele and one increased-functional allele (RMs) or two increased-functional alleles of CYP2C19 (UMs).
  Interventions: Drug: Control session; Drug: Inhibition session; Drug: Induction session

INTERVENTIONS:
Drug: Control session — Plasma and urine sampling as well as the determination of the blood OH-omeprazole/omeprazole ratio at baseline by capillary blood sampling.
Drug: Inhibition session — Plasma and urine sampling as well as the determination of the blood OH-omeprazole/omeprazole ratio at baseline by capillary blood sampling, with prior administration of 50 mg of fluvoxamine for 7 consecutive days (CYP2C19 inhibitor).
Drug: Induction session — Plasma and urine sampling as well as the determination of the blood OH-omeprazole/omeprazole ratio at baseline by capillary blood sampling, with prior administration of 600 mg of rifampicin for 10 consecutive days (CYP2C19 inducer).

SUMMARY:
The objective of this clinical trial is to identify endogenous compounds (substances naturally present in the human body) that may serve as predictors of the activity of a key liver enzyme, CYP2C19. This enzyme plays a crucial role in the metabolism of several important drugs and exhibits significant interindividual variability in its activity, which can contribute to adverse drug reactions or reduced therapeutic efficacy.

The study will involve 40 healthy volunteers, divided into two groups: 10 poor metabolizers and 30 non-poor metabolizers. Each participant will undergo three sessions.

In the first session, 24-hour urine collection and plasma sampling will be conducted. Omeprazole will be administered orally, and the baseline blood OH-omeprazole/omeprazole ratio will be determined via capillary blood sampling.

The second session, identical in procedure to the first, will take place after 7 days of fluvoxamine administration (inhibition phase). The third session will also mirror the first but will follow 10 days of rifampicin administration (induction phase).

Endogenous compounds showing significant variation across sessions and between metabolizer groups will be evaluated as potential biomarkers for predicting CYP2C19 activity.

DETAILED DESCRIPTION:
CYP2C19 is involved in the metabolism of approximately 6.8% of all marketed drugs. Its enzymatic activity varies significantly between individuals due to genetic polymorphisms, environmental factors, ethnicity, or disease states. While the administration of a CYP2C19 probe drug, such as omeprazole, is a reliable method for phenotyping this enzyme, it is relatively invasive and not suitable for certain vulnerable populations, such as pregnant women.

Identifying an endogenous compound metabolized by CYP2C19 could provide a non-invasive alternative to conventional phenotyping methods. This clinical study aims to identify such endogenous biomarkers by evaluating the effects of genetic variation, enzyme inhibition and induction on the metabolome of healthy volunteers.

To achieve this, untargeted metabolomic profiling using ultra-high-performance liquid chromatography coupled with high-resolution mass spectrometry (UHPLC-HRMS) will be conducted on plasma, extracellular vesicles and urine samples.

This single-centre, open-label clinical trial will enroll 40 healthy participants (both men and women), aged 18 to 65 years. Participants will be assigned to one of two groups based on their CYP2C19 genotype: poor metabolizers (PMs) and normal, rapid, or ultrarapid metabolizers (NMs, RMs, UMs).

Each participant will undergo three study sessions:

Session 1: CYP2C19 phenotyping following a single 10 mg oral dose of omeprazole.

Session 2: Identical to Session 1, but following a 7-day pretreatment with fluvoxamine (CYP2C19 inhibitor, 50 mg once daily).

Session 3: Identical to Session 1, but following a 10-day pretreatment with rifampicin (CYP2C19 inducer, 600 mg once daily).

In all sessions, urine will be collected for 24 hours and venous blood samples will be taken prior to omeprazole administration for metabolomics analysis. Capillary blood will also be sampled after omeprazole intake to assess the CYP2C19 phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Age 18-65 years
* Body Mass Index (BMI) 18-27
* Understanding of French language and able to give a written inform consent
* CYP2C19 genotype: PMs, NMs, RMs or UMs
* At least one barrier method contraception during the whole study and 1 month after the end of the study (in addition of hormonal contraception if applicable)

Exclusion Criteria:

* CYP2C19 IMs
* Participation in any other interventional clinical study within 3 months prior to inclusion
* Pregnant or breastfeeding woman
* Any pathologies, use of drugs or food that may affect CYP activity (based on the 'drug interactions and cytochromes P450 table published by the Service of Clinical Pharmacology and Toxicology, HUG50 and on the investigator's knowledge)
* Medical history of liver transplantation
* Regular smokers of ≥ 10 cigarettes/day
* Alcohol intake 2 days prior to session 1 and during fluvoxamine and rifampicin intake
* Alteration of hepatic tests (ASAT, ALAT, GGT, bilirubin more than 3x normal)
* Renal failure (serum urea, serum creatinine and eGFR outside the norms)
* Medical history of chronic alcoholism or abuse of psychoactive drugs
* Sensitivity to any of the drugs used
* Psychiatric disorders
* Beck Score ≥10 (question related to suicide >0)
* Contact lens wearers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Fold-change in the intensities of features determined by mass spectrometry according to genotype (PMs versus NMs-RMs-UMs) and according to sessions. | Samples collected at Session 1 (Day 1), Session 2 (Day 11 ± 4), and Session 3 (Day 27 ± 4); data analysis completed within 90 days after the final session of the last participant.
  Metabolic features showing a fold-change ≥ 1.5 or ≤ 0.6737 will be qualified as CYP2C19 endogenous biomarkers. Chromatographic signals will be detected in healthy volunteers' urine, plasma and liver-derived extracellular vesicles by liquid chromatography coupled to high resolution mass spectrometry (LC-HRMS) at each session for each volunteer.

SECONDARY OUTCOMES:
Correlation of significant ions measured in metabolomics with OH-OPZ/OPZ blood ratio. | Within 90 days after the last study session of the last participant.
Predictive performance metrics of a multivariate linear regression model for CYP2C19 phenotype. | Within 90 days after the last study session of the last participant.

CONTACTS AND LOCATIONS:
Locations (1):
- The Geneva University Hospitals (HUG), Geneva, Switzerland

DOCUMENTS (1):
  • Study Protocol (2024-08-09): https://cdn.clinicaltrials.gov/large-docs/30/NCT07014930/Prot_000.pdf